CLINICAL TRIAL: NCT01407068
Title: An Open-label Study to Assess the Safety and Efficacy of Concurrent Administration of Two Injections of AA4500 0.58 mg Into the Same Hand of Subjects With Multiple Dupuytren's Contractures
Brief Title: Administration of Two Injections for Multiple Dupuytren's Contractures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-864
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Results first posted 2015-02-20 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Dupuytren's Contracture
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AA4500 (Experimental): AA4500 collagenase clostridium histolyticum
  Interventions: Biological: AA4500 collagenase clostridium histolyticum

INTERVENTIONS:
Biological: AA4500 collagenase clostridium histolyticum — 2 concurrent injections (0.58 mg) into 2 cords on the same hand
  Other Names: Xiaflex; Xiapex

SUMMARY:
The objectives of this study are to assess the safety and efficacy of concurrent administration of two injections of AA4500 into the same hand of subjects with multiple Dupuytren's contractures caused by palpable cords.

DETAILED DESCRIPTION:
Methodology/Study Design:

This is an open-label, study in men and women with multiple Dupuytren's contractures. Approximately 60 subjects who have at least two Dupuytren's contractures caused by palpable cords in the same hand will be enrolled.

After all pre-injection procedures are completed on Day 1, eligible men and women will receive two concurrent injections of AA4500 0.58 mg into the same hand. On Day 2, a finger extension procedure to facilitate cord disruption will be performed in those subjects who do not have spontaneous disruption of their cord(s). Follow-up visits for the evaluation of safety and efficacy will be on Day 8, Day 30, and Day 60.

Upon completion of the Day 60 follow-up visit, subjects who require further treatment will have the option to receive three additional open-label treatments according to the XIAFLEX package insert (Appendix C). Subjects may receive up to a total of five injections and individual cords may receive up to a total of three injections.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Be a man or woman ≥ 18 years of age
3. Have a diagnosis of Dupuytren's disease and have at least 2 fixed-flexion contractures on the same hand that are ≥ 20º in PIP and/or MP joints in fingers, other than the thumbs, which are caused by palpable cords suitable for treatment
4. Have a positive "table top test" defined as the inability to simultaneously place the affected finger(s) and palm flat against a table top
5. Either be using an accepted method of birth control (ie, surgical sterilization; intra uterine contraceptive device; oral contraceptive; diaphragm or condom in combination with contraceptive cream, or jelly or foam) and have negative pregnancy testing before administration of AA4500, if a female of childbearing potential, or be a postmenopausal female (no menses for at least 1 year or hysterectomy)
6. Not have any clinically significant medical history or condition(s) that would, in the opinion of the investigator, substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives of the study
7. Be able to comply with the study visit schedule as specified in the protocol

Exclusion Criteria:

1. Received surgery (fasciectomy or surgical fasciotomy) and/or needle aponeurotomy/fasciotomy on the selected joints to be treated within 90 days before the first injection of AA4500
2. Has a chronic muscular, neurological, or neuromuscular disorder that affects the hands
3. Has a known systemic allergy to collagenase or any other excipient of AA4500
4. Has received any collagenase treatments (eg, Santyl® ointment and/or XIAFLEX/XIAPEX) within 30 days before injection of AA4500
5. Is currently receiving or plans to receive anticoagulant medication or has received anticoagulant medication (except for ≤ 150 mg aspirin daily and over-the-counter nonsteroidal anti-inflammatory drugs [NSAIDs]) within 7 days before injection of AA4500)
6. Has a known recent history of stroke, bleeding, or other medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
7. Is known to be immunocompromised or human immunodeficiency virus (HIV) positive
8. Has a history of illicit drug abuse or alcoholism within the year before injection of AA4500
9. Received an investigational drug within 30 days before injection of AA4500
10. Is a pregnant or lactating female
11. Has any clinically significant medical history or condition(s), including conditions that affect the hands, that would, in the opinion of the investigator, substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives of the study
12. Has jewelry on the hand to be treated that cannot be removed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD, MPPH, Study Director — Endo Pharmaceuticals
Locations (7):
- United States (4):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - The Indiana Hand Center, Indianapolis, Indiana
  - Department of Orthopaedics SUNY-Stony Brook, Stony Brook, New York
  - Health Research Institute, Oklahoma City, Oklahoma
- Australia (3):
  - AusTrials, Auchenflower
  - AusTrials, Kippa-Ring
  - Emeritus Research, Malvern

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AA4500
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AA4500
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 21
  Australia | 39

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Fixed Flexion
Description: Total fixed flexion is defined as the sum of the fixed flexion contractures of the two joints receiving treatment. Change in fixed-flexion contracture is measured in degrees where a decrease of 100% would correspond to a reduction in contracture to 0 degrees
Time Frame: 30 days after last injection
Population: Efficacy analysis is based of the intent-to-treat population (ITT). The population is defined as all enrolled subjects who received two injections of AA4500 and had at least one-post-injection measurement.
Measure: Mean (Standard Deviation); unit: percentage of contracture change
Arm/Group | AA4500
Number analyzed (Participants) | 60
percentage of contracture change | 75.5 (24.11)

2. Secondary Outcome: Subject Satisfaction With Treatment
Description: At the Day 60 follow-up visit, each subject will be asked to rate his/her satisfaction with treatment as follows:
  1. Very Satisfied
  2. Quite Satisfied
  3. Neither Satisfied nor Dissatisfied
  4. Quite Dissatisfied
  5. Very Dissatisfied
Time Frame: 60 days after last injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AA4500
Number analyzed (Participants) | 60
participants
  Very satisfied | 36
  Quite satisfied | 17
  Neither satisfied nor dissatisfied | 5
  Quite dissatisfied | 1
  Very dissatisfied | 1
  Not done | 0

3. Secondary Outcome: Investigator Assessment of Improvement With Treatment
Description: At the Day 60 follow-up visit, the investigator will determine the degree of improvement in the severity of the subject's treated finger(s) compared with screening as follows:
  1. Very Much Improved
  2. Much improved
  3. Minimally Improved
  4. No Change
  5. Minimally Worse
  6. Much Worse
  7. Very Much Worse
Time Frame: 60 days after last injection
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AA4500
Number analyzed (Participants) | 60
participants
  Very much improved | 33
  Much improved | 22
  Minimally improved | 4
  No change | 1
  Minimally worse | 0
  Much worse | 0
  Very much worse | 0
  Not done | 0

4. Primary Outcome: Change in Total Range of Motion
Description: The total range of motion is the sum of the range of motion measurements of the two treated joints. Range of motion is defined as difference between full flexion angle and full extension angle expressed in degrees.
Time Frame: 30 days after last injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | AA4500
Number analyzed (Participants) | 60
degrees | 60.4 (21.80)

5. Secondary Outcome: Clinical Success by Joint Type
Description: Clinical success is defined as a reduction in fixed flexion contracture to 5° or less 30 days after injection of AA4500.
Time Frame: 30 days after injection
Population: as for outcome 1
Measure: Number; unit: number of joints
Units Other Than Participants: Number of joints
Groups:
- AA4500 MP: AA4500 collagenase clostridium histolyticum
  AA4500 collagenase clostridium histolyticum: 2 concurrent injections (0.58 mg) into 2 cords on the same hand in the metacarpophalangeal (MP) joint cord
- AA4500 PIP: AA4500 collagenase clostridium histolyticum
  AA4500 collagenase clostridium histolyticum: 2 concurrent injections (0.58 mg) into 2 cords on the same hand in the interphalangeal (PIP) joint cord
Arm/Group | AA4500 MP | AA4500 PIP
Number analyzed (Participants) | 60 | 60
Number analyzed (Number of joints) | 75 | 45
number of joints
  Yes | 57 | 15
  No | 18 | 30

ADVERSE EVENTS:
Time Frame: 60 days after injection
Arm/Group | AA4500
Serious Adverse Events (participants affected / at risk) | 3/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=60)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=60)
oedema peripheral (General disorders) | 49 (53)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 (53)
Contusion (Injury, poisoning and procedural complications) | 48 (55)
Lymphadenopathy (Blood and lymphatic system disorders) | 22 (23)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (20)
Skin laceration (Injury, poisoning and procedural complications) | 15 (16)
Injection site haematoma (General disorders) | 11 (14)
Injection site swelling (General disorders) | 8 (9)
Blood blister (Skin and subcutaneous tissue disorders) | 7 (7)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other